CLINICAL TRIAL: NCT01969968
Title: Lipophilic Organic Polluants and Morbid Obesity: Kinetic of the Release and Impact on the Metabolic Syndrome Before and After Bariatric Surgery
Brief Title: Lipophilic Organic Polluants and Morbid Obesity
Acronym: POLOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-API-01
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- sleeve bariatric surgery (Other): morbidly obese adults, with or without metabolic syndrome eligible for bariatric surgery undergoing sleeve gastrectomy
  Interventions: Other: Lipophilic Organic Polluants dosage
- morbidly obese adults with by pass surgery (Other): morbidly obese adults, with or without metabolic syndrome eligible for bariatric surgery undergoing gastric bypass
  Interventions: Other: Lipophilic Organic Polluants dosage
- non obese (Other): non obese patients
  Interventions: Other: Lipophilic Organic Polluants dosage

INTERVENTIONS:
Other: Lipophilic Organic Polluants dosage — Urinary, blood and fat dosage of Lipophilic Organic Polluants

SUMMARY:
1. To study the kinetics of release after bariatric surgery of selected polluants stored in adipose tissue, looking for clinical and/or predictive factors
2. To test the hypothesis of a deleterious effect of this release on the expected improvement of insulin-resistance and on the liver inflammation.
3. To determine the level of contamination of morbidly obese patients, with or without metabolic syndrome, compared to a control, non obese population, with special attention to clinical (age, gender, reproductive history, pregnancy, nursing) and biological parameters (insulin-resistance, inflammation).

DETAILED DESCRIPTION:
I- Goals Because of its exponential prevalence and its co-morbidities, obesity, particularly in its most massive forms, has become a public health problem. It is likely that this epidemic be secondary to both genetic and behavioural factors, and also to environmental factors. Specifically, the "obesogen" and "diabetogen" role of several persistant organic polluants (POP) known as endocrine disruptors used in farming or industry has recently been suggested by experimental animal studies and by human epidemiologic studies. Those chemicals are usually lipophilic, are stored in adipose tissue where they bio-accumulate, and are released in the blood stream during the lipolysis that occurs in any weight loss. This weight loss is particularly rapid and important after bariatric surgery, that is proposed as a treatment for morbid obesity usually leading to an improvement of insulin resistance, metabolic syndrome, and diabetes. However, this improvement is not constant, or is less important than would be anticipated for the massive weight loss observed. This raises the question of the importance and of deleterious impact of the blood release of lipophilic POPs on the evolution of metabolic syndrome and the low grade associated inflammation.

In a prospective, multicentric study, we propose to analyse the kinetic of the release of several POPs during rapid and massive weight loss obtained after bariatric surgery. Those POPs have been chosen for their obesogen or diabetogen properties, reported in vitro or in vivo, for their lipophilic nature, and their ubiquitous presence in the home environment and/or into the food chain: bisphenol A (plastics); tributyltin (fungicide, anti-fouling agent or thermic stabilizant); polybrominated diphenyl ethers (PBDE, fire retardants); perchlorated octanoïd acid and its sulphated compounds (PFOA and PFOS, perfluoroalkyls used as surfactant, lubrifiants, and usted in wrappings); and organochorinated compounds such as: PCB153, representing the polychlorinated bisphenyls (electric isolation); hexachlorobenzene (HBC), and several pesticides: DDE, metabolite of DDT, now banned but with a very long half life, hexachlorocyclohexane (HCH), heptachlor, nanochlor and chlordane used in agriculture.

II- Originality and /or new aspect of the project Though suggested by several experimental studies, the role of POP in human obesity remains largely unknown.

There are no or very few papers on the role in humans of the POPs we have selected, but they are supported by animal experimental studies.

The concept of release in the blood stream after weight loss is recent and deserves to be studied.

III- Reasons for the choice of questions (3 maximum) Interest of the results/method to improve knowledge on those questions

1. To study the kinetics of release after bariatric surgery of selected polluants stored in adipose tissue, looking for clinical and/or predictive factors
2. To test the hypothesis of a deleterious effect of this release on the expected improvement of insulin-resistance and on the liver inflammation.
3. To determine the level of contamination of morbidly obese patients, with or without metabolic syndrome, compared to a control, non obese population, with special attention to clinical (age, gender, reproductive history, pregnancy, nursing) and biological parameters (insulin-resistance, inflammation).

IV- Description of the methods/ Calendar The POPs will be measured in serum, urine (for BPA) and in adipose tissue (subcutaneous and visceral) by gas chromatography coupled to mass spectrometry.

Fat mass will be estimated when possible by DEXA (if weight<150 kg), or by impedancemetry, allowing the calculation of an estimated total body burden for each POP (since they are lipophilic, we will multiply the concentration of each chemical in adipose tissue expressed in ng/g of fat by the total estimated body mass of fat).

The number of patients included will be 250 morbidly obese adults, with or without metabolic syndrome (3 out of 5 classical criteria), eligible for bariatric surgery (125 from Nice undergoing gastric bypass, and 125 from Montpellier undergoing sleeve gastrectomy).

Concentrations of polluants will be measured at baseline and 3, 6 and 12 month after bariatric surgery, and at 18 months as well for patients who will undergo abdominoplasty required by their massive weight loss. Baseline concentrations in obese patients will be compared to those measured in 100 controls, matched for age and gender, with a BMI<25.

Insulin resistance will be assessed by HOMA-IR, adiponectine and SHBG, inflammation by us CRP, leptin, interleukin 6, TNF alpha, transaminases, gammaGT, alkalin phosphatase.

The redistribution of POPs in serum and adipose tissue, and the estimation of total body burden will be assessed before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* health coverage
* mentally competent
* signed consent form
* stable weight over the last three months

Non inclusion criteria :

* pregnancy
* insulin treated diabetes
* significant weight change over the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
measurement of POPs | 18 months
  Urinary and blood POPs dosage 18 months after bariatric surgery
clinical and biological assessment of metabolic syndrome | 18 months after bariatric surgery
  blood dosage for clinical and biological assessment of metabolic syndrome including glucose tolerance test 18 months after bariatric surgery

SECONDARY OUTCOMES:
Kinetic profiles of POP release within 18 months following bariatric surgery | 18 months following bariatric surgery
  blood and urinary dosage
Total body burden of selected POPs before and after surgery | before surgery and 18 months after surgery
  Total body burden of selected POPs before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick FENICHEL, PhD, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Nice, France